CLINICAL TRIAL: NCT01155921
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Dr.Reddy's Laboratories Ltd. and Janssen Pharmaceutica Products, LP. (Risperdal M-TABTM)1 mg Risperidone Orally Disintegrating Tablets in Healthy Adult Male Volunteers Under Fasting Conditions
Brief Title: Bioavailability Study of Risperidone Orally Disintegrating Tablets 1 mg of Dr.Reddy's Laboratories Limited Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Vice President, Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA19885
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioavailability; Crossover; Risperidone
MeSH Terms: interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone Orally Disintegrating (Experimental): Risperidone Orally Disintegrating Tablets 1 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Risperidone Orally Disintegrating Tablets
- Risperdal M-TAB (Active Comparator): (Risperdal M-TAB) 1 mg risperidone orally disintegrating tablets Janssen Pharmaceutica Products
  Interventions: Drug: Risperidone Orally Disintegrating Tablets

INTERVENTIONS:
Drug: Risperidone Orally Disintegrating Tablets — Risperidone Orally Disintegrating Tablets 1 mg of Dr.Reddy's Laboratories Limited
  Other Names: (Risperdal M-TAB) tablets of Janssen Pharmaceutica Products

SUMMARY:
The purpose of this study was to assess the single-dose relative bioavailability study of 1 mg risperidone orally disintegrating tablets and (Risperdal M-TAB) under fasting conditions.

DETAILED DESCRIPTION:
Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Dr Reddy's Laboratories Ltd. and Janssen Pharmaceutica Products, LP. (Risperdal M-TAB) 1 mg Risperidone Orally Disintegrating Tablets in Healthy Adult Male Volunteers under Fasting Conditions

ELIGIBILITY:
Inclusion Criteria:

Subjects were included in the study only if they met all of the following criteria:

* Healthy non-smoking (for at least 3 months) adult male volunteers, 18-45 years of age;
* Weighing at least 60 kg for males and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983);
* Medically healthy subjects with clinically normal laboratory profiles and ECGs;
* Voluntarily consent to participate in the study.

Exclusion Criteria:

Subjects were excluded from the study if there was evidence of any of the following at screening or at any time during the study:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic,neurologic, or psychiatric disease.
* In addition, history or presence of:
* alcoholism or drug abuse within the past year;
* hypersensitivity or idiosyncratic reaction to risperidone or benzodiazepines or other antipsychotic drugs;
* seizures;
* glaucoma or hypermetropia.
* Positive results on Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HbsAg) and Hepatitis C Virus (HCV) Tests.
* Subjects whose sitting blood pressure is less than 110/60 mm Hg at screening or 100/55 mm Hg before dosing.
* Subjects whose pulse is lower than 55 b.p.m. at screening or 50 b.p.m. prior to dosing. Subjects whose PR interval is ≥ 190 msec at screening and prior to dosing.
* Subjects whose aTe interval is > 450 msec at screening and prior to dosing.
* Subjects with a body temperature ≥38°C before dosing.
* Subjects who have used any drugs or substances known to be strong inhibitors of CYP enzymes (formerly known as cytochrome P450 enzymes) within 10 days prior to the first dose.
* Subjects who have used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
* Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who, through completion of the study, would have donated in excess of: 500 mL of blood in 14 days, or 1500 mL of blood in 180 days, 2500 mL of blood in 1 year.
* Subjects who have participated in another clinical trial within 28 days prior to the first dose.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2004-08; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Bioavailability based on Cmax and AUC parameters | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Geatano Morelli, M.D, Principal Investigator — MDS Pharma Services